CLINICAL TRIAL: NCT06198179
Title: Effects of Upper Limb Children Action-observation Training (UP-CAT) With and Without Visual Feedback in Children With Cerebral Palsy
Brief Title: Effects of UP-CAT With and Without Visual Feedback in Children With CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0753
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy (CP),; Rehabilitation; Upper extremity; Activities of daily living
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: This study will be randomized controlled trial (RCT) used to measure the effects of upper limb action-observation training (UP-CAT) with and without visual feedback in children with cerebral palsy. subjects with cerebral palsy meeting pre determined inclusion and exclusion criteria will be be divided into two groups using non-probability sampling techniques.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): these individuals will receive the upper limb children action-observation training (UP-CAT) with visual feedback
  UP-CAT:
  * Individual tasks like modelling compound,board games,cards,magnets,glass bead to do bracelets,painting and crafting (making a grass man,making musical instruments with cardboard),cooking (making juice cocktails,fruit skewers,chocolate fondue),building towers, making puzzles & water games including filling a bucket with a sponge/bottle,filling & throwing water balloons.
  * To maximize the variety of the actions we included different objects (e.g.coins,bottles, stamps,modelling compound) to be grasped with different grasp types (whole hand,pinch, tripod grasp) and in different orientations of the wrist.
  Visual feedback:
  Mirror in front of patient will be used. After the baseline assessment,the patient in the experimental group will receive the upper limb children action-observation training with visual feedback Time of rehabilitation will be 1 hour/subject.
  Interventions: Other: upper limb children action-observation training (UP-CAT) with visual feedback
- Control group (Other): This will receive the upper limb children action-observation training (UP-CAT).
  UP-CAT:
  Following tasks will be performed by children
  * Individual tasks like modelling compound,board games,cards,magnets,glass bead to do bracelets,painting and crafting (making a grass man,making musical instruments with cardboard),cooking (making juice cocktails,fruit skewers,chocolate fondue),building towers, making puzzles & water games including filling a bucket with a sponge/bottle,filling & throwing water balloons
  * To maximize the variety of the actions we included different objects (e.g. coins,bottles, stamps,modelling compound) to be grasped with different grasp types (whole hand,pinch, tripod grasp) & in different orientations of the wrist.After the baseline assessment,the patient in the experimental group will receive the UL children action-observation training with visual feedback Time of rehabilitation will be 1 hour per subject.
  Interventions: Other: upper limb children action-observation training (UPCAT)

INTERVENTIONS:
Other: upper limb children action-observation training (UPCAT) — upper limb children action-observation training (UPCAT) without visual Feedback
  Arms: Control group
Other: upper limb children action-observation training (UP-CAT) with visual feedback — upper limb children action-observation training (UP-CAT) with visual feedback: Mirror therapy as visual feedback
  Arms: Experimental group

SUMMARY:
Cerebral palsy (CP) is the most common neurological disorder of movement and/or posture and of motor function, which are due to a non-progressive interference or abnormality of the developing brain. In hemiplegic cerebral palsy (HCP), one side of the body is involved with the upper extremity more affected than the lower. HCP is treated by addressing the underlying cause and by various form of therapy to recover motor function. Motor function in hemi paretic limb particularly fine motor skill may be improved by upper limb children action-observation therapy (UP-CAT).

DETAILED DESCRIPTION:
This will be randomized controlled trial. Non-probability purposive sampling technique will be used for recruiting samples for study. Children will be assessed by House Functional Classification System for hemiplegia to include in the study. Computerized randomization will be used to locate subjects in two groups, and 28 hemiplegic cerebral palsy children will be divided into 2 groups; experimental and control groups. In experimental group hemiplegic cerebral palsy children will perform upper limb exercises with visual feedback for 5 times a week, 15 sets of daily life upper limb activities, each action will be observed for 2 minutes and executed for 2 minutes. In control group hemiplegic cerebral palsy children will perform upper limb activities for 5 times a week, 15 sets of daily life upper limb activities, each action will be observed for 2 minutes and executed for 2 minutes. Both groups will be assessed at the time of recruitment and at the end of 4 weeks. Data will be collected by Melbourne unilateral upper limb (MUUL) and ABILHAND-kids questionnaire. After collection of data, data will be analyzed by SPSS-25.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy children aged 5 years to 10 years at the time of recruitment.
* Both male and female
* According to Modified Ashworth scale of spasticity; score should be +1.
* Mild or moderate UL disability i.e. active use of affected UL from poor active assist use to complete spontaneous use according to House Functional Classification System grade between 4 and 8.

Exclusion Criteria:

* Individuals with the other neurological deficits
* Visual impairment.
* Children with upper limb disabilities other than hemiplegic cerebral palsy.
* Children with uncontrolled epileptic seizures in last 3 years
* Non co-operative patients.
* Previous orthopedic surgery or botulinum toxin A (BoNT-A) injection in the UL within 6 months prior to the enrolment of this study.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Melbourne Assessment of Unilateral Upper Limb Function (MUUL) | 4 weeks
  The MUUL is an evaluative tool that measures unilateral upper extremity quality of movement in children with neurological impairments aged from 5 to 15 years. MUUL is a criterion-referenced test based on 16 items scored on a 3- to 5-point ordinal scale comprising tasks that are representative of the most important components of unilateral UL function
ABILHAND-Kids | 4 weeks
  The ABILHAND-Kids is a short questionnaire that measures 21 mainly bimanual daily activities referred to the activity domain of the ICF. The difficulty experienced by the child to perform the required tasks is scored by a parent on a 3-point ordinal scale (impossible, difficult, and easy).

CONTACTS AND LOCATIONS:
Overall Officials: IQRA Muhammad Afzal, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sgandurra G, Cecchi F, Beani E, Mannari I, Maselli M, Falotico FP, Inguaggiato E, Perazza S, Sicola E, Feys H, Klingels K, Ferrari A, Dario P, Boyd RN, Cioni G. Tele-UPCAT: study protocol of a randomised controlled trial of a home-based Tele-monitored UPper limb Children Action observation Training for participants with unilateral cerebral palsy. BMJ Open. 2018 May 14;8(5):e017819. doi: 10.1136/bmjopen-2017-017819. PMID 29764869